CLINICAL TRIAL: NCT05546450
Title: Determination of the Effect of Lyophilized Dried Cornus Mas L. Fruit Powder on Nutritional Status in Individuals With Metabolic Associated Fatty Liver Disease Combined With Medical Nutrition Therapy
Brief Title: Effect of Lyophilized Cornus Mas L. on Anthropometric and Biochemical Parameters in Metabolic Associated Fatty Liver Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Hatice Merve Bayram, Principal Investigator (Assist. Prof.), Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2019.810
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Fatty Liver Disease; Obesity; Liver Fat
Keywords: Metabolic associated fatty liver disease; Cornus mas L.; diet treatment; nutrition therapy; anthropometric measurements
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Fatty Liver | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Group (No Intervention): Among those who applied to the clinic, those who do not want to follow their diet will be randomized into this group.
- Cornus mas L. and Diet Group (Experimental): Among those who applied to the clinic, those who want to follow their diet will be randomized into this group. Patients in this group will be followed by a personalized diet and will receive 30 g/day lyophilized Cornus mas L. fruit powder for their one portion of fruit a day.
  Interventions: Behavioral: Diet; Dietary Supplement: Cornus mas L.(Cornelian Cherry)
- Diet Group (Experimental): Among those who applied to the clinic, those who want to follow their diet will be randomized into this group. Patients in this group will be followed by a personalized diet.
  Interventions: Behavioral: Diet
- Cornus mas L. Group (Experimental): Among those who applied to the clinic, those who do not want to follow their diet will be randomized into this group. Patients in this group will receive 30 g/day lyophilized Cornus mas L. fruit powder
  Interventions: Dietary Supplement: Cornus mas L.(Cornelian Cherry)
- Healthy Control Group (No Intervention): This group included healthy individuals who were not diagnosed with Metabolic Associated Fatty Liver.

INTERVENTIONS:
Behavioral: Diet — Patient in "Diet Group" and "Cornus mas L. and Diet Group" will be given a personalized diet and be followed up by a dietician.
  Arms: Cornus mas L. and Diet Group; Diet Group
Dietary Supplement: Cornus mas L.(Cornelian Cherry) — Patients in "Cornus mas L. Group" and "Cornus mas L. and Diet Group" will receive 30 g/day freeze-dried Cornus mas L. fruit powder supplement.
  Arms: Cornus mas L. Group; Cornus mas L. and Diet Group

SUMMARY:
The aim of the study was to evaluate the effect of lyophilized Cornus mas L. fruit powder with/without diet therapy on biochemical parameters and anthropometric measurements in patients with metabolic associated fatty liver disease.

DETAILED DESCRIPTION:
The main purpose of this study is to determine the efficacy of the lyophilized dried powder form of cornelian cherry (Cornus mas L.) grown in our country on nutritional status and biochemical parameters in patients with metabolic-associated fatty liver disease.

Sub-objectives of the study;

* Determination of the effect of cornelian cherry on blood glucose, and lipid parameters, and liver enzymes.
* Determination of anti-inflammatory, antidiabetic, and antioxidant effects of cornelian cherry in metabolic fatty liver patients.
* Determination of the effect of cornelian cherry on anthropometric measurements.

The aim of this study is to compare the anthropometric measurements and biomarkers of patients with metabolic-associated fatty liver disease as a result of the consumption of powdered cornelian cherry (Cornus mas L.) that has been freeze-dried at -55 degrees with a Lyophilizer device for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years with metabolic associated fatty liver.
* Those who applied to the gastroenterology clinic
* Volunteers
* Those who signed the consent form

Exclusion Criteria:

* Those with <18 to ≥65 years
* Those without ultrasonography results
* Those with >20 g/day for men and 10 g/day for women alcohol consumption in the past 1 year
* Those with hepatitis B or C
* Those with chronic liver diseases associated with viral hepatitis, such as Wilson disease, hemochromatosis, and Cushing syndrome
* Those with autoimmune liver disease
* Those with a history of cardiovascular diseases, cancer, mental diseases, severe liver, and kidney dysfunction
* Those with thyroid diseases such as goiter, hypothyroidism, or hyperthyroidism
* Those with prolonged use of estrogen or regular consumption of drugs associated with fatty liver diseases, such as corticosteroid, methotrexate, tamoxifen, and amiodarone
* Pregnant, breastfeeding women
* Those with allergic to Cornus mas fruit
* Those with an unwillingness to continue the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting blood glucose (mg/dL) at 8 weeks | 8 weeks
  The fasting blood glucose at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in blood lipid parameters (mg/dL) at 8 weeks | 8 weeks
  The total triglyceride, cholesterol, LDL, and HDL at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in Aspartate transaminase (AST) (u/L) at 8 weeks | 8 weeks
  The AST levels at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in BMI (kg/m2) at 8 weeks | 8 weeks
  The body weight (kg) and height (m) of the patients with metabolic-associated fatty liver disease will be taken every 15 days for 8 weeks by trained and qualified nutritionists using standardized procedures and noted in their files. Height will be measured to the nearest 0.1 cm using a stadiometer, with shoes off. Tanita SC-330 (Accurate Technology Co., Ltd. Tianjin, China) was used to analyze body composition, and the subjects' body weight, percentage of lean mass, and fat were recorded. Body mass index (BMI) will be calculated as weight (kg) divided by height (m) squared.
Change from baseline in fasting insulin (mU/L) at 8 weeks | 8 weeks
  The fasting insulin at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in HOMA-IR at 8 weeks | 8 weeks
  The HOMA-IR at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in hbA1c (%) at 8 weeks | 8 weeks
  The hbA1c at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in Alanine Transaminase (ALT) (u/L) at 8 weeks | 8 weeks
  The ALT at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in Gamma-Glutamyl Transpeptidase (GGT) (u/L) at 8 weeks | 8 weeks
  The GGT at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in Alkaline phosphatase (ALP) (u/L) at 8 weeks | 8 weeks
  The ALP at the baseline and 8 weeks later will be taken noted from the routinely requested tests in the hospital. These values will be recorded for all groups; Control Group, the Diet Group (who received a diet for 8 weeks), Cornelian Cherry and Diet Group (who received an additional 30 g/day of dried powdered Cornelian Cherry with their diet), Cornelian Cherry Group (who was given only 30 g/day of dried powdered Cornelian Cherry ), and Healthy Control Group.
Change from baseline in circumference measurements (meters) at 8 weeks | 8 weeks
  Circumference measurements will be taken every 15 days for 8 weeks by trained and qualified nutritionists using standardized procedures.These measurements are; waist circumference (cm), hip circumference(cm), mid-upper arm circumference(cm), neck circumference(cm), waist to height ratio(cm) and waist to hip ratio(cm).
  Circumferences will be measured using a non-stretch plastic tape measure with an accuracy of 1 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Merve Bayram, phD, Principal Investigator — Istanbul Gelisim University
Locations (1):
- Istanbul Gelisim University, Istanbul, Avcılar, Turkey (Türkiye)